CLINICAL TRIAL: NCT03274687
Title: A Randomized Phase III Trial of Hypofractionated Post-Prostatectomy Radiation Therapy (HYPORT) Versus Conventional Post-Prostatectomy Radiation Therapy (COPORT)
Brief Title: Hypofractionated Radiation Therapy or Conventional Radiation Therapy After Surgery in Treating Patients With Prostate Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GU003; NCI-2016-01771 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GU003; NRG-GU003 (Other: NRG Oncology); NRG-GU003 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Results first posted 2022-06-06 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Prostate Adenocarcinoma; Stage I Prostate Adenocarcinoma AJCC v7; Stage II Prostate Adenocarcinoma AJCC v7; Stage III Prostate Adenocarcinoma AJCC v7
MeSH Terms: interventions — Radiation Dose Hypofractionation; Radiation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (conventional radiation therapy) (Experimental): Patients undergo conventional radiation therapy for 37 fractions over 7 weeks in the absence of disease progression or unacceptable toxicity. Patients may also receive androgen deprivation therapy for up to 6 months as per doctor recommendation.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy
- Arm II (hypofractionated radiation therapy (Experimental): Patients undergo hypofractionated radiation therapy for 25 fractions over 5 weeks in the absence of disease progression or unacceptable toxicity. Patients may also receive androgen deprivation therapy for up to 6 months as per doctor recommendation.
  Interventions: Radiation: Hypofractionated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated; Hypofractionated Radiotherapy; hypofractionation; Radiation, Hypofractionated
  Arms: Arm II (hypofractionated radiation therapy
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo conventional radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Arm I (conventional radiation therapy)

SUMMARY:
This randomized phase III trial studies how well hypofractionated radiation therapy works compared to conventional radiation therapy after surgery in treating patients with prostate cancer. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects. Conventional radiation therapy uses high energy x-rays, gamma rays, neutrons, protons, or other sources to kill tumor cells and shrink tumors. It is not yet known whether giving hypofractionated radiation therapy or conventional radiation therapy after surgery may work better in treating patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate that hypofractionated post-prostatectomy radiotherapy (HYPORT) does not increase patient-reported gastrointestinal (GI) or genitourinary (GU) symptoms over conventionally fractionated post-prostatectomy (COPORT) at the 2-year time point.

SECONDARY OBJECTIVES:

I. To compare patient-reported GI symptoms using the Expanded Prostate Cancer Index Composite (EPIC)-26 at end of radiation therapy (RT) and 6, 12, 24, and 60 months from end of treatment.

II. To compare patient-reported GU symptoms using the EPIC-26 at end of RT and 6, 12, 24, and 60 months from end of treatment.

III. To compare time to progression (TTP) where progression is defined as the first occurrence of biochemical failure (BF), local failure, regional failure, distant metastasis (DM), institution of new unplanned anticancer treatment, or death from prostate cancer (prostate cancer specific mortality [PCSM]).

IV. To compare freedom from biochemical failure (FFBF) and TTP rates with an alternate prostate specific antigen (PSA) >= PSA nadir + 2 ng/mL definition of BF.

V. To compare local failure, regional failure, salvage therapy (i.e. institution of new unplanned anticancer treatment), DM, PCSM, and overall survival (OS) rates.

VI. Assessment of adverse events.

EXPLORATORY OBJECTIVES:

I. To compare utilities for health outcomes using the EuroQol five dimensions questionnaire (EQ-5D).

II. Paraffin-embedded tissue block, serum, plasma, whole blood, and urine for future translational research analyses for predictors of toxicity following hypofractionated or conventionally fractionated post-prostatectomy radiotherapy.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo conventional radiation therapy for 37 fractions over 7 weeks in the absence of disease progression or unacceptable toxicity. Patients may also receive androgen deprivation therapy for up to 6 months as per doctor recommendation.

ARM II: Patients undergo hypofractionated radiation therapy for 25 fractions over 5 weeks in the absence of disease progression or unacceptable toxicity. Patients may also receive androgen deprivation therapy for up to 6 months as per doctor recommendation.

After completion of study treatment, patients are followed up every 6 months for 2 years and every year for 3 years and thereafter.

ELIGIBILITY:
Inclusion Criteria:

* PRIOR TO STEP 1 REGISTRATION
* Adenocarcinoma of the prostate treated primarily with radical prostatectomy

  * Any type of radical prostatectomy will be permitted, including retropubic, perineal, laparoscopic, or robotically assisted; there is no time limit for the date of radical prostatectomy
* One of the following pathologic T-classifications: pT2 or pT3

  * Patients with positive surgical margins are eligible
* One of the following pathologic N-classifications: pN0, pNX

  * If a lymph node dissection is performed, the number of lymph nodes removed per side of the pelvis and the extent of the pelvic lymph node dissection (obturator versus [vs.] extended lymph node dissection) should be noted whenever possible
* No clinical evidence of regional lymph node metastasis

  * Computed tomography (CT) (with contrast if renal function is acceptable; a noncontrast CT is permitted if the patient is not a candidate for contrast), magnetic resonance imaging (MRI), nodal sampling, or dissection of the pelvis within 120 days prior to step 1 registration
  * Patients with pelvic lymph nodes equivocal or questionable by imaging are eligible if the nodes are =< 1 cm in the short axis
* A post-radical prostatectomy study entry PSA >= 45 days after prostatectomy and within 30 days prior to step 1, < 2.0 ng/mL
* No evidence of a local recurrence in the prostate fossa based on a digital rectal examination (DRE) within 60 days prior to step 1 registration

  * Patients with equivocal or questionable DRE findings should have an MRI of the pelvis to exclude the presence of a prostate fossa mass
  * Patients with equivocal or questionable exam findings by DRE or MRI are eligible if a biopsy of the lesion is negative for tumor
* No evidence of bone metastases (M0) on bone scan (Na F positron emission tomography (PET)/CT is an acceptable substitute) within 120 days prior to step 1 registration

  * Equivocal bone scan findings are allowed if plain films and/or MRI are negative for metastasis
* Zubrod performance status 0-1 within 60 days prior to step 1 registration
* The patient or a legally authorized representative must provide study-specific informed consent prior to step 1 registration
* Willingness and ability to complete the Expanded Prostate Cancer Index Composite (EPIC) questionnaire
* Only English and French-speaking patients are eligible to participate as these are the only language the EPIC has been validated in
* PRIOR TO STEP 2 REGISTRATION
* The EPIC must be completed in full and entered within 10 business days after step 1 registration; NRG Oncology Statistical and Data Management Center has 3 business days to score the results and send a notification to the site to proceed to step 2 randomization

Exclusion Criteria:

* A post-prostatectomy PSA nadir >= 0.2 ng/mL AND Gleason >= 7 (Considered for NRG-GU002, principal investigator [PI]: Hurwitz)
* pT2 with a negative surgical margin and PSA < 0.1 ng/mL
* Androgen deprivation therapy started prior to prostatectomy for > 6 months (180 days) duration;

  * Note: The use of finasteride or dutasteride (+/- tamsulosin) for longer periods prior to prostatectomy is acceptable
* Androgen deprivation therapy started after prostatectomy and prior to step 1 registration for > 6 weeks (42 days)
* Neoadjuvant chemotherapy before or after prostatectomy
* Prior invasive (except non-melanoma skin cancer) malignancy unless disease-free for a minimum of 3 years and not in the pelvis; (for example, carcinoma in situ of the oral cavity is permissible if disease free for a minimum of 3 years; however, patients with prior history of bladder cancer are not allowed no matter the disease free duration); prior hematological (e.g., leukemia, lymphoma, myeloma) malignancy is not allowed
* Previous chemotherapy for any other disease site if given within 3 years prior to step 1
* Prior radiotherapy, including brachytherapy, to the region of the study cancer that would result in overlap of radiation therapy treatment volumes
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of step 1 registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of step 1 registration
  * Severe hepatic disease, defined as a diagnosis of Child-Pugh class B or C hepatic disease
  * Human immunodeficiency virus (HIV) positive with cluster of differentiation (CD)4 count < 200 cells/microliter; note that patients who are HIV positive are eligible, provided they are under treatment with highly active antiretroviral therapy (HAART) and have a CD4 count >= 200 cells/microliter within 30 days prior to registration; note also that HIV testing is not required for eligibility for this protocol
  * End-stage renal disease (ie, on dialysis or dialysis has been recommended)
* Prior allergic reaction to the study drugs involved in this protocol
* History of inflammatory bowel disease, prior bowel surgeries (or colostomy) for any reason, or prior partial/radical cystectomy for any reason

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2026-08-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mark K Buyyounouski, Principal Investigator — NRG Oncology
Locations (241):
- United States (229):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Marin Cancer Care Inc, Greenbrae, California
  - Marin General Hospital, Greenbrae, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Yale University, New Haven, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - SIH Cancer Institute, Carterville, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Goshen Center for Cancer Care, Goshen, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - East Jefferson General Hospital, Metairie, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - University of Maryland Radiation Oncology Center at Union Hospital, Elkton, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Beth Israel Deaconess Hospital-Plymouth, Plymouth, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Michigan Healthcare Professionals Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan Healthcare Professionals Farmington, Farmington Hills, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - McLaren Cancer Institute-Owosso, Owosso, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Michigan Healthcare Professionals Troy, Troy, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Lovelace Radiation Oncology, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - UNC Health Cancer Care Raleigh, Raleigh, North Carolina
  - Novant Cancer Institute Radiation Oncology - Supply, Supply, North Carolina
  - Novant Health Cancer Institute Radiation Oncology - Wilmington, Wilmington, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic Akron General, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Crozer-Keystone Regional Cancer Center at Broomall, Broomall, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Crozer Regional Cancer Center at Brinton Lake, Glen Mills, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - The Radiation Oncology Center-Hilton Head/Bluffton, Hilton Head Island, South Carolina
  - Carolina Regional Cancer Center, Myrtle Beach, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Farmington Health Center, Farmington, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Ogden Regional Medical Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Overlake Medical Center, Bellevue, Washington
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Mayo Clinic Health System Eau Claire Hospital-Luther Campus, Eau Claire, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Canada (11):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Centre De Sante Et De Services Sociaux De Chicoutimi, Chicoutimi, Quebec
  - CIUSSSEMTL-Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Kantonsspital Aarau, Aarau, Switzerland

REFERENCES:
- [Derived] Buyyounouski MK, Pugh SL, Chen RC, Mann MJ, Kudchadker RJ, Konski AA, Mian OY, Michalski JM, Vigneault E, Valicenti RK, Barkati M, Lawton CAF, Potters L, Monitto DC, Kittel JA, Schroeder TM, Hannan R, Duncan CE, Rodgers JP, Feng F, Sandler HM. Noninferiority of Hypofractionated vs Conventional Postprostatectomy Radiotherapy for Genitourinary and Gastrointestinal Symptoms: The NRG-GU003 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2024 May 1;10(5):584-591. doi: 10.1001/jamaoncol.2023.7291. Erratum In: JAMA Oncol. 2024 Jun 1;10(6):833. doi: 10.1001/jamaoncol.2024.1062. JAMA Oncol. 2025 Dec 1;11(12):1555. doi: 10.1001/jamaoncol.2025.4707. PMID 38483412

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 298 screened, 296 participants were randomized.
Groups:
- Conventional Radiation Therapy: Conventional post-prostatectomy radiation therapy (COPORT) over 7 weeks. Patients may also receive optional androgen deprivation therapy per doctor recommendation.
  Conventional radiation therapy: 66.6 Gy in 37 daily fractions of 1.8 Gy to the prostate bed in the absence of disease progression or unacceptable toxicity.
  Optional androgen deprivation therapy (ADT): Any luteinizing hormone-releasing hormone (LHRH) agonist/antagonist with or without an oral antiandrogen can be used up to a six-month administration dose, starting 7-9 weeks before radiation therapy and may begin as early as 42 days prior to or any time after screening. An oral antiandrogen alone is not allowed.
- Hypofractionated Radiation Therapy: Hypofractionated post-prostatectomy radiation therapy (HYPORT) over 5 weeks. Patients may also receive optional androgen deprivation therapy per doctor recommendation.
  Hypofractionated radiation therapy: 62.5 Gy in 25 daily fractions of 2.5 Gy to the prostate bed in the absence of disease progression or unacceptable toxicity.
  Optional androgen deprivation therapy: Any LHRH agonist/antagonist with or without an oral antiandrogen can be used up to a six-month administration dose, starting 7-9 weeks before radiation therapy and may begin as early as 42 days prior to or any time after screening. An oral antiandrogen alone is not allowed.
Period: Overall Study
Arm/Group | Conventional Radiation Therapy | Hypofractionated Radiation Therapy
Started | 152 | 144
Eligible | 151 | 143
Eligible With Adverse Event Data | 148 | 141
Completed (Participants contributing data to results are considered to have completed the study.) | 151 | 143
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: Eligible participants
Groups:
- Conventional Radiation Therapy: Conventional post-prostatectomy radiation therapy (COPORT) over 7 weeks. Patients may also receive optional androgen deprivation therapy per doctor recommendation.
  Conventional radiation therapy: 66.6 Gy in 37 daily fractions of 1.8 Gy to the prostate bed in the absence of disease progression or unacceptable toxicity.
  Optional androgen deprivation therapy: Any LHRH agonist/antagonist with or without an oral antiandrogen can be used up to a six-month administration dose, starting 7-9 weeks before radiation therapy and may begin as early as 42 days prior to or any time after screening. An oral antiandrogen alone is not allowed.
- Total: Total of all reporting groups
Arm/Group | Conventional Radiation Therapy | Hypofractionated Radiation Therapy | Total
Number analyzed (Participants) | 151 | 143 | 294
Age, Customized [Count of Participants; unit: Participants] — Years
  Participants
    ≤ 49 years | 3 | 2 | 5
    50 - 59 years | 27 | 31 | 58
    60 - 69 years | 74 | 83 | 157
    ≥ 70 years | 47 | 27 | 74
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 151 | 143 | 294
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 142 | 136 | 278
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 21 | 43
  White | 125 | 114 | 239
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
EPIC Group [Count of Participants; unit: Participants] — The EPIC is a prostate cancer health-related quality of life (HRQOL) self-administered instrument measuring patient-reported urinary, bowel, sexual, and hormonal symptoms related to prostate cancer treatments. Response options for each item form a Likert scale with scores transformed linearly to a 0-100 scale. Domain scores are also on a 0-100 scale with higher scores representing better HRQOL. The urinary domain contains 12 items. The bowel domain contains 14 items.
  Participants
    A Score Group (bowel domain score > 96, urinary domain score > 84) | 56 | 52 | 108
    B Score Group (bowel domain score > 96, urinary domain score ≤ 84) | 29 | 32 | 61
    C Score Group (bowel domain score ≤ 96, urinary domain score > 84) | 31 | 31 | 62
    D Score Group (bowel domain score ≤ 96, urinary domain score ≤ 84) | 35 | 28 | 63
Prior androgen deprivation therapy (ADT) [Count of Participants; unit: Participants]
  No | 118 | 110 | 228
  Yes | 33 | 33 | 66
Prostate-specific antigen (PSA) ng/mL [Count of Participants; unit: Participants] — Prostate-specific antigen (PSA) is a protein made by the prostate gland and found in the blood. PSA blood levels may be higher than normal in men who have prostate cancer, benign prostatic hyperplasia (BPH), or infection or inflammation of the prostate gland, and are often used to monitor patients who have been treated for prostate cancer to see if their cancer has recurred.
  Participants
    0.0 - 0.5 | 135 | 128 | 263
    0.6 - 1.0 | 10 | 14 | 24
    1.1 - 1.5 | 3 | 1 | 4
    1.6 - 2.0 | 3 | 0 | 3
Gleason score [Count of Participants; unit: Participants] — Gleason score describes prostate cancer based on how abnormal the cancer cells in a biopsy sample look under a microscope. Cells are scored 1-5 with 1 indicating "low-grade" looking similar to normal cells and 5 indicating "high-grade" barely resembling normal cells due to mutation. A pathologist assigns a Gleason grade to the first and second most predominant patterns in the biopsy. The two grades are added together to calculate the Gleason score (between 2 and 10). Cancers with lower scores tend to be less aggressive, while cancers with higher scores end to be more aggressive.
  Participants
    6 | 16 | 7 | 23
    7 | 105 | 109 | 214
    8 | 14 | 15 | 29
    9 | 15 | 11 | 26
    10 | 1 | 1 | 2
T-Stage [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) 7th ed. refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues.
  Participants
    T2 | 76 | 60 | 136
    T3 | 75 | 83 | 158
N-Stage [Count of Participants; unit: Participants] — Regional lymph nodes staging per American Joint Committee on Cancer (AJCC) refers to the number and/or extent of spread of lymph nodes that contain cancer. A higher number means the cancer is in more lymph nodes, farther away from the original tumor. N0 means lymph nodes aren't involved; NX means the lymph nodes could not be assessed.
  Participants
    NX | 30 | 33 | 63
    N0 | 121 | 110 | 231
Zubrod [Count of Participants; unit: Participants] — 0 = Asymptomatic; 1 = Symptomatic but completely ambulatory; 2 = Symptomatic, <50% in bed during the day; 3 = Symptomatic, >50% in bed, but not bedbound; 4 = Bedbound; 5 = Death
  Participants
    0 | 128 | 127 | 255
    1 | 23 | 16 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change in Urinary Domain of the Expanded Prostate Cancer Index (EPIC) at Two Years
Description: The EPIC is a prostate cancer health-related quality of life (HRQOL) self-administered instrument measuring patient-reported urinary, bowel, sexual, and hormonal symptoms related to prostate cancer treatments. Response options for each item form a Likert scale with scores transformed linearly to a 0-100 scale. Domain scores are also on a 0-100 scale with higher scores representing better HRQOL. The urinary domain contains 12 items. Change from baseline is calculated by subtracting baseline from later score, with a positive change score indicating increased HRQOL.
Time Frame: Baseline (randomization), 2 years
Population: Eligible participants with baseline and two-year data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Radiation Therapy | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 127 | 117
units on a scale | -4.12 (14.72) | -5.06 (15.16)
Statistical Analysis 1: Comparison: Conventional Radiation Therapy vs Hypofractionated Radiation Therapy; Null hypothesis (H0): mean change score of HYPORT (∆2) is worse than that of COPORT (∆1), specifically ∆2 - ∆1 < -5. Alternative hypothesis (HA): ∆2 is not worse than ∆1, specifically ∆2 - ∆1 ≥ -5. The study sample size is based on 90% power for this endpoint and 91% power for the bowel endpoint (resulting in 81.9% statistical power to reject the null hypothesis for both endpoints) and a one-sided alpha=0.025 with an overall type I error of 0.05 with a Bonferroni adjustment; Test type: Non-Inferiority — The non-inferiority margin for the difference in mean change score (∆2 - ∆1) is -5; p = 0.98, t-test, 1 sided

2. Primary Outcome: Change in Bowel Domain of the Expanded Prostate Cancer Index (EPIC) at Two Years
Description: The EPIC is a prostate cancer health-related quality of life (HRQOL) self-administered instrument measuring patient-reported urinary, bowel, sexual, and hormonal symptoms related to prostate cancer treatments. Response options for each item form a Likert scale with scores transformed linearly to a 0-100 scale. Domain scores are also on a 0-100 scale with higher scores representing better HRQOL. The bowel domain contains 14 items. Change from baseline is calculated by subtracting baseline from later score, with a positive change score indicating increased HRQOL.
Time Frame: Baseline, 2 years
Population: Eligible participants with baseline and two-year data
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Conventional Radiation Therapy | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 127 | 117
units on a scale | -1.42 (8.35) | -4.21 (11.0)
Statistical Analysis 1: Comparison: Conventional Radiation Therapy vs Hypofractionated Radiation Therapy; Null hypothesis (H0): mean change score of HYPORT (∆2) is worse than that of COPORT (∆1), specifically ∆2 - ∆1 < -5. Alternative hypothesis (HA): ∆2 is not worse than ∆1, specifically ∆2 - ∆1 ≥ -5. The study sample size is based on 91% power for this endpoint and 90% power for the urinary endpoint (resulting in 81.9% statistical power to reject the null hypothesis for both endpoints) and a one-sided alpha=0.025 with an overall type I error of 0.05 with a Bonferroni adjustment; Test type: Non-Inferiority — The non-inferiority margin for the difference in mean change score (∆2 - ∆1) is -6; p = 0.96, t-test, 1 sided

3. Secondary Outcome: Change in Urinary Domain Score of the Expanded Prostate Cancer Index (EPIC) at End of Radiation Therapy (RT), 6 Months, 1 and 5 Years
Description: as for outcome 1
Time Frame: Baseline, end of RT, then 6 months,1 and 5 years from the start of RT (5 year time point has not yet been reached). RT dates depend on timing and duration of androgen deprivation therapy (ADT) (optional) and RT.
Population: Eligible participants with baseline data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Radiation Therapy | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 151 | 143
units on a scale
  End of RT | -4.34 (22.61) | -7.90 (20.93)
  6 months | 0.08 (20.26) | -1.71 (18.55)
  1 year | -2.32 (22.63) | -5.41 (21.15)
Statistical Analysis 1: Comparison: Conventional Radiation Therapy vs Hypofractionated Radiation Therapy; End of RT; Test type: Superiority; p = 0.70, t-test, 2 sided
Statistical Analysis 2: Comparison: Conventional Radiation Therapy vs Hypofractionated Radiation Therapy; 6 months; Test type: Superiority; p = 0.67, t-test, 2 sided
Statistical Analysis 3: Comparison: Conventional Radiation Therapy vs Hypofractionated Radiation Therapy; 1 year; Test type: Superiority; p = 0.66, t-test, 2 sided

4. Secondary Outcome: Change in Bowel Domain Score of the Expanded Prostate Cancer Index (EPIC) at End of RT, 6 Months, 1 and 5 Years
Description: as for outcome 2
Time Frame: Baseline, end of RT, then 6 months,1 and 5 years from the start of RT (5 year time point has not yet been reached). RT dates depend on timing and duration of ADT (optional) and RT.
Population: Eligible participants with baseline data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Radiation Therapy | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 151 | 143
units on a scale
  End of RT | -6.83 (15.82) | -14.96 (21.32)
  6 months | -1.90 (13.63) | -2.70 (13.98)
  1 year | -2.67 (12.65) | -3.11 (13.93)
Statistical Analysis 1: Comparison: Conventional Radiation Therapy vs Hypofractionated Radiation Therapy; End of RT; Test type: Superiority; p = 0.0011, t-test, 2 sided
Statistical Analysis 2: Comparison: Conventional Radiation Therapy vs Hypofractionated Radiation Therapy; 6 months; Test type: Superiority; p = 0.93, t-test, 2 sided
Statistical Analysis 3: Comparison: Conventional Radiation Therapy vs Hypofractionated Radiation Therapy; 1 year; Test type: Superiority; p = 0.30, t-test, 2 sided

5. Secondary Outcome: Percentage of Participants With Biochemical Failure
Description: Biochemical failure was analyzed using two different definitions. The protocol definition of biochemical failure is a PSA measurement ≥ 0.4 ng/mL and rising (i.e. PSA ≥ 0.4 ng/mL followed by a value higher than the first by any amount) or followed by initiation of salvage hormones. The Phoenix definition of biochemical failure is a PSA measurement ≥ PSA nadir + 2 ng/mL where nadir is the lowest post-RT PSA value. Time to biochemical failure is defined as time from randomization to the date of first biochemical failure, last known follow-up (censored), or death without biochemical failure (competing risk). Biochemical failure rates are estimated using the cumulative incidence method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Two-year rates are provided.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 3.0 years.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conventional Radiation Therapy | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 151 | 143
percentage of participants
  Protocol definition | 8.3 [4.5 to 13.6] | 11.8 [7.0 to 17.9]
  Phoenix definition | 3.5 [1.3 to 7.4] | 8.0 [4.2 to 13.3]
Statistical Analysis 1: Comparison: Conventional Radiation Therapy vs Hypofractionated Radiation Therapy; Protocol definition of biochemical failure; Test type: Superiority; p = 0.29, Gray's test; Two-sided significance level 0.05
Statistical Analysis 2: Comparison: Conventional Radiation Therapy vs Hypofractionated Radiation Therapy; Phoenix definition of biochemical failure; Test type: Superiority; p = 0.22, Gray's test; Two-sided significance level 0.05

6. Secondary Outcome: Percentage of Participants With Progression
Description: Progression (failure) is defined as the first occurrence of biochemical failure, local failure, regional failure, distant failure, institution of new unplanned anticancer treatment, or death from prostate cancer. Time to progression is defined as time from randomization to the date of progression, last known follow-up (censored), or death without progression (competing risk). Progression rates are estimated using the cumulative incidence method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Two-year rates are provided.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 3.0 years. Two-year rates reported here. Follow-up schedule: end of RT, then 6, 12, 18, 24 months from start of RT, then yearly.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conventional Radiation Therapy | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 151 | 143
percentage of participants | 14.4 [9.3 to 20.6] | 14.7 [9.3 to 21.2]
Statistical Analysis 1: Comparison: Conventional Radiation Therapy vs Hypofractionated Radiation Therapy; Test type: Superiority; p = 0.96, Gray's test — Two-sided significance level 0.05

7. Secondary Outcome: Percentage of Participants With Local-Regional Failure
Description: Local-regional failure is defined as local or regional failure. Local failure is defined as the development of a new biopsy-proven mass in the prostate bed. Regional failure is defined as radiographic evidence (CT or MRI) of lymphadenopathy (lymph node size ≥ 1.0 cm in the short axis) in a patient without the diagnosis of a hematologic/lymphomatous disorder associated with adenopathy. Time to local-regional failure is defined as time from randomization to the date of first local-regional failure, last known follow-up (censored), or death without local-regional (competing risk). Local-regional failure rates are estimated using the cumulative incidence method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Two-year rates are provided.
Time Frame: as for outcome 6
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conventional Radiation Therapy | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 151 | 143
percentage of participants | 0.7 [0.1 to 3.5] | 0.8 [0.1 to 3.8]
Statistical Analysis 1: Comparison: Conventional Radiation Therapy vs Hypofractionated Radiation Therapy; Test type: Superiority; p = 0.35, Gray's test — Two-sided significance level 0.05

8. Secondary Outcome: Percentage of Participants Receiving Salvage Therapy
Description: Salvage therapy is defined as the initiation of new unplanned anticancer treatment. Time to salvage therapy initiation is defined as time from randomization to the date of first salvage therapy, last known follow-up (censored), or death without salvage therapy (competing risk). Salvage therapy rates are estimated using the cumulative incidence method. The protocol specifies that the distributions of salvage initiation times be compared between the arms, which is reported in the statistical analysis results. Two-year rates are provided.
Time Frame: as for outcome 6
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conventional Radiation Therapy | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 151 | 143
percentage of participants | 7.5 [3.9 to 12.5] | 5.8 [2.7 to 10.6]
Statistical Analysis 1: Comparison: Conventional Radiation Therapy vs Hypofractionated Radiation Therapy; Test type: Superiority; p = 0.41, Gray's test — Two-sided significance level 0.05

9. Secondary Outcome: Percentage of Participants With Distant Metastasis
Description: Distant metastasis (failure) is defined as radiographic evidence of hematogenous spread evaluated by bone scan, CT, or MRI. Time to distant metastasis is defined as time from randomization to the date of first distant metastasis, last known follow-up (censored), or death without local recurrence (competing risk). Distant metastasis rates are estimated using the cumulative incidence method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Two-year rates are provided.
Time Frame: as for outcome 6
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conventional Radiation Therapy | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 151 | 143
percentage of participants | 0.7 [0.1 to 3.5] | 2.2 [0.6 to 5.8]
Statistical Analysis 1: Comparison: Conventional Radiation Therapy vs Hypofractionated Radiation Therapy; Test type: Superiority; p = 0.60, Gray's test — Two-sided significance level 0.05

10. Secondary Outcome: Percentage of Participants Who Died From Prostate Cancer (Prostate Cancer Specific Mortality)
Description: Cause of death was centrally reviewed. Count and percentage at time of analysis are reported.
Time Frame: as for outcome 6
Population: Eligible participants
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Radiation Therapy | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 151 | 143
Participants | 0 | 0

11. Secondary Outcome: Percent of Participants Alive (Overall Survival)
Description: Overall survival time is defined as time from registration/randomization to the date of death (failure) from any cause or last known follow-up (censored). Overall survival rates are estimated by the Kaplan-Meier method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. 2-year rates are provided.
Time Frame: as for outcome 6
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conventional Radiation Therapy | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 151 | 143
percentage of participants | 98.6 [97.0 to 100.0] | 98.5 [96.8 to 100.0]
Statistical Analysis 1: Comparison: Conventional Radiation Therapy vs Hypofractionated Radiation Therapy; Test type: Superiority; p = 0.61, Log Rank — Two-side significance level 0.05; Hazard Ratio (HR) = 1.58, 95% CI 2-sided [0.26 to 9.47] — Reference = COPORT

12. Secondary Outcome: Number of Participants With Grade 3+ Adverse Events
Description: Common Terminology Criteria for Adverse Events (CTCAE) version 4 grades adverse event severity from 1=mild to 5=death. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data. Counts of participants with any grade 3 or higher adverse event, any grade 3 or higher gastrointestinal adverse events, and any grade 3 or higher genitourinary adverse events are reported. Adverse events of any attribution are included.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 3.0 years. Follow-up schedule: end of RT, then 6, 12, 18, 24 months from start of RT, then yearly.
Population: Eligible with adverse event data
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Radiation Therapy | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 148 | 141
Participants
  All adverse events | 25 | 20
  Gastrointestinal Adverse Events | 3 | 2
  Genitourinary Adverse Events | 6 | 10
Statistical Analysis 1: Comparison: Conventional Radiation Therapy vs Hypofractionated Radiation Therapy; Patients with any grade 3 or higher adverse event of any attribution; Test type: Superiority; p = 0.53, Chi-squared
Statistical Analysis 2: Comparison: Conventional Radiation Therapy vs Hypofractionated Radiation Therapy; Patients with any grade 3 or higher gastrointestinal adverse event of any attribution; Test type: Superiority; p = 0.6929, Chi-squared
Statistical Analysis 3: Comparison: Conventional Radiation Therapy vs Hypofractionated Radiation Therapy; Patients with any grade 3 or higher genitourinary adverse event of any attribution; Test type: Superiority; p = 0.2605, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events were to be evaluated at end of RT, then every 6 months from start of RT for two years, then yearly. RT dates depends on timing and duration of ADT (optional) and RT. Maximum follow-up at time of of analysis was 3.0 years.
Description: All-cause mortality was assessed in eligible participants. Adverse events were assessed in eligible participants with adverse event data.
Arm/Group | Conventional Radiation Therapy | Hypofractionated Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/143
Serious Adverse Events (participants affected / at risk) | 1/148 | 8/141
Other Adverse Events (participants affected / at risk) | 130/148 | 120/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conventional Radiation Therapy (N=148) | Hypofractionated Radiation Therapy (N=141)
Myocardial infarction (Cardiac disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Anaphylaxis (Immune system disorders) | 0 | 1
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 3
Hematuria (Renal and urinary disorders) | 0 | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 1
Renal calculi (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Conventional Radiation Therapy (N=148) | Hypofractionated Radiation Therapy (N=141)
Abdominal pain (Gastrointestinal disorders) | 8 | 5
Constipation (Gastrointestinal disorders) | 17 | 17
Diarrhea (Gastrointestinal disorders) | 43 | 53
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 13 | 17
Proctitis (Gastrointestinal disorders) | 8 | 18
Rectal hemorrhage (Gastrointestinal disorders) | 6 | 18
Fatigue (General disorders) | 80 | 62
Urinary tract infection (Infections and infestations) | 8 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 7
Cystitis noninfective (Renal and urinary disorders) | 12 | 10
Hematuria (Renal and urinary disorders) | 9 | 20
Renal and urinary disorders - Other (Renal and urinary disorders) | 36 | 22
Urinary frequency (Renal and urinary disorders) | 75 | 73
Urinary incontinence (Renal and urinary disorders) | 45 | 48
Urinary retention (Renal and urinary disorders) | 14 | 9
Urinary tract pain (Renal and urinary disorders) | 11 | 15
Urinary urgency (Renal and urinary disorders) | 43 | 45
Erectile dysfunction (Reproductive system and breast disorders) | 24 | 18
Hot flashes (Vascular disorders) | 37 | 32
Hypertension (Vascular disorders) | 8 | 11

LIMITATIONS AND CAVEATS:
Local and regional failure data was collected as a combined event (local-regional progression) and therefore is reported as a single outcome measure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/87/NCT03274687/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/87/NCT03274687/ICF_001.pdf